CLINICAL TRIAL: NCT06244290
Title: : Clinical Study to Assess the Efficacy of a Dentifrice Containing Stannous Fluoride as Compared to a Commercially-available Potassium-based Toothpaste and a Regular Fluoride Toothpaste (Negative Control) on the Reduction of Dentinal Hypersensitivity.
Brief Title: Dentinal Hypersensitivity Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2020-05-SEN-SNF-CA-BGS
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Dentinal Hypersensitivity
Keywords: tactile; airblast; dentin hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Centers for Disease Control and Prevention, U.S.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (Active Comparator): Colgate SnF Toothpaste Colgate Adult Extra Clean soft-bristle toothbrush
  Interventions: Drug: Colgate SNF; Drug: Sensodyne Extra Whitening; Drug: Colgate Fluoride (CDC)
- Group II (Active Comparator): Sensodyne Extra Whitening Toothpaste Colgate Adult Extra Clean soft-bristle toothbrush
  Interventions: Drug: Colgate SNF; Drug: Sensodyne Extra Whitening; Drug: Colgate Fluoride (CDC)
- Group III (Placebo Comparator): Colgate Fluoride Toothpaste (CDC) Colgate Adult Extra Clean soft-bristle toothbrush
  Interventions: Drug: Colgate SNF; Drug: Sensodyne Extra Whitening; Drug: Colgate Fluoride (CDC)

INTERVENTIONS:
Drug: Colgate SNF — toothpaste
Drug: Sensodyne Extra Whitening — toothpaste
Drug: Colgate Fluoride (CDC) — toothpaste

SUMMARY:
The objective of this clinical study is to assess the efficacy of a dentifrice containing stannous fluoride (Colgate-Palmolive Company, New York, NY, USA) as compared to a commercially-available potassium-based toothpaste (Sensodyne Extra Whitening Toothpaste, GlaxoSmithKline Co., UK) and a commercially available non-desensitizing toothpaste (Colgate Cavity Protection Toothpaste, Colgate-Palmolive Company, New York, NY, USA) in the reduction of dentinal hypersensitivity over a seven (7) day period.

ELIGIBILITY:
Inclusion Criteria:

* Sign an Informed Consent Form;
* Male or female 18 to 70 years of age, inclusive;
* Be in good general health as determined by the study investigators;
* Available for the seven (7) days duration of the study;
* Must present two (2) sensitive teeth which must meet ALL of the following criteria:

  * Be anterior to the molars and demonstrating dentin exposure due to cervical erosion/abrasion and/or gingival recession;
  * Have a qualifying dentin hypersensitivity response to tactile stimuli applied to the cervical surface (gingivo-facial 1/3) as defined by a response score between 10- 50grams of force (Yeaple Probe, XiniX Research Inc. Portsmouth, NH, USA);
  * Have a qualifying dentin hypersensitivity response to air blast stimuli applied for one second to the cervical surface (gingivo-facial 1/3) as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale

Exclusion Criteria:

* Gross oral pathology, chronic disease, and/or history of allergies to any of the test products;
* Use of a desensitizing oral care product and/or recipient of any dental desensitizing treatment within the past three months prior to start of the study;
* Advanced periodontal disease and/or treatment for periodontal disease (including surgery) within the past twelve months;
* Sensitive teeth with a mobility greater than one;
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures;
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily use of analgesics;
* Participation in any other oral clinical study for the duration of this study
* Self-reported pregnancy and/or currently breastfeeding;
* Allergies to oral care products, personal care consumer products, and/or their ingredients;
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Tactile dentin hypersensitivity | Baseline, 1-Day, 3-Days and 7-Days
  Have a qualifying dentin hypersensitivity response to tactile stimuli applied to the cervical surface (gingivo-facial 1/3) as defined by a response score between 10- 50grams of force (Yeaple Probe, XiniX Research Inc. Portsmouth, NH, USA)
Air blast dentin hypersensitivity | Baseline, 1-Day, 3-Days and 7-Days
  Have a qualifying dentin hypersensitivity response to air blast stimuli applied for one second to the cervical surface (gingivo-facial 1/3) as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Farid Ayad, DMD, MSD, Principal Investigator — Mesa Dental Centre
Locations (1):
- Mesa Dental Centre, Costa Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No